CLINICAL TRIAL: NCT05721859
Title: Medacta M-Vizion™ Macroscopic Radiographic Study, Multi-center, Post-Market Outcomes Study
Brief Title: M-Vizion™ Macroscopic Radiographic Study
Status: Recruiting | Type: Observational
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: MUSA-H-MV-001
Record Dates: First submitted 2023-01-27; First posted 2023-02-10 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Revision Hip Arthroplasty
Keywords: revision; hip; arthroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: revision hip arthroplasty — revision hip arthroplasty

SUMMARY:
Study of the patient's subsidence after revision hip arthroplasty by assessing gross stem subsidence in the femoral canal.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the M-Vizion modular stem performance in patients who undergo total hip replacement according to the standard practice. It is expected that subjects receiving revision hip arthroplasty with the Medacta M-Vizion™ modular hip stem will have less than 5mm of stem subsidence at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read, understand, and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF).
* Ability to understand and provide written authorization for use and disclosure of personal health information.
* Subjects who are able and willing to comply with the study protocol and follow-up visits.
* Patients requiring a revision total hip replacement.
* Subjects undergoing revision THA who will receive an M-Vizion femoral component according to the indications for use.
* Male and female patients ages 21 - 80 years of age at the time of surgery.

Exclusion Criteria:

* Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* Patients with a systemic or metabolic disorder leading to progressive bone deterioration.
* Patients bone stock is compromised by disease or infection, which could possibly prevent adequate support and/or fixation to the prosthesis.
* Patients with an active or suspected latent infection in or about the hip joint.
* Patients that are incarcerated.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for revision THA receiving a M-Vizion femoral component and meeting all inclusion/ exclusion criteria at a research site,
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
subsidence | 6 weeks post-op visit (± 2 weeks)
  Occurrence of subsidence >5mm
subsidence | 6 Months post-op visit (± 2 months)
  Occurrence of subsidence >5mm
subsidence | 1 year post-op visit (± 4 months)
  Occurrence of subsidence >5mm
subsidence | 2 year post-op visit (± 6 months)
  Occurrence of subsidence >5mm

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Northwestern Medicine, Chicago, Illinois
  - New England Baptist Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth Health, Lebanon, New Hampshire
  - OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Utah Department of Orthopaedics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No